CLINICAL TRIAL: NCT04026555
Title: Realtime Streaming Clinical Use Engine for Medical Escalation
Acronym: ReSCUE-ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Matthew Levin, Associate Professor, Department of Anesthesiology, Perioperative & Pain Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 19-0729
Record Dates: First submitted 2019-07-16; First posted 2019-07-19 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Clinical Deterioration; Hospital Medicine; Monitoring, Physiologic
Keywords: Medical Early Warning Systems; Patient Monitoring; Electronic Health Record; Big Data; Critical Care; Machine Learning
MeSH Terms: conditions — Clinical Deterioration

STUDY DESIGN:
Intervention Model Description: For each patient, real-time data from clinical and administrative systems will be used by ReSCUE-ME to produce a MEWS++ score predicting the likelihood that the patient will require escalation of care within the next 6 hours. Upon the patient being admitted to the unit, the patient will be evaluated based on any update in the EHR. If the prediction score exceeds a "high" threshold, the RRT team will be notified directly. If the score is between a "low" threshold and the high threshold , the nursing team will be notified and increased nursing monitoring will be initiated. If the patient has met criteria for increased nursing monitoring, a refractory 8-hour refractory window will be applied during which no nursing alerts will be sent. However if the score exceeds the high threshold, the RRT team will be notified. Throughout the trial, the performance of the alerts will be monitored via web-based dashboards. If the performance is poor, the "high" and "low" thresholds will be adjusted.
Masking Description: No masking is completed as the information/waiver of consent sheet for the two arms needed to be individualized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEWS++ Monitoring (Active Comparator): This consists of all the patients that will be receiving MEWS++ escalation monitoring and provider alerting.
  Interventions: Other: MEWS++ Monitoring; Other: Predictor Score
- Standard of Care Monitoring (Placebo Comparator): Patients in the control arm will have a score calculated but no alert will be sent.
  Interventions: Other: Predictor Score

INTERVENTIONS:
Other: MEWS++ Monitoring — Patient's electronic medical record data will undergo processing by a machine learning algorithm (MEWS++).
  Arms: MEWS++ Monitoring
Other: Predictor Score — A score predicting the likelihood that the patient will experience a deterioration in their clinical condition within six hours will be generated. If the prediction score exceeds a predetermined threshold, an alert will be sent to the provider. The alerting protocol is tiered, with both a low and high threshold. If the score is above the low threshold, nursing will be notified. If the score is above the high threshold, RRT will be notified.

SUMMARY:
The escalation of care for patients in a hospitalized setting between nurse practitioner managed services, teaching services, step-down units, and intensive care units is critical for appropriate care for any patient. Often such "triggers" for escalation are initiated based on the nursing evaluation of the patient, followed by physician history and physical exam, then augmented based on laboratory values. These "triggers" can enhance the care of patients without increasing the workload of responder teams. One of the goals in hospital medicine is the earlier identification of patients that require an escalation of care. The study team developed a model through a retrospective analysis of the historical data from the Mount Sinai Data Warehouse (MSDW), which can provide machine learning based triggers for escalation of care (Approved by: IRB-18-00581). This model is called "Medical Early Warning Score ++" (MEWS ++). This IRB seeks to prospectively validate the developed model through a pragmatic clinical trial of using these alerts to trigger an evaluation for appropriateness of escalation of care on two general inpatients wards, one medical and one surgical. These alerts will not change the standard of care. They will simply suggest to the care team that the patient should be further evaluated without specifying a subsequent specific course of action. In other words, these alerts in themselves does not designate any change to the care provider's clinical standard of care. The study team estimates that this study would require the evaluation of ~ 18380 bed movements and approximately 30 months to complete, based on the rate of escalation of care and rate of bed movements in the selected units.

DETAILED DESCRIPTION:
Objectives:

Mount Sinai Hospital has developed a Rapid Response Team (RRT) system designed to give general floor care providers additional support for patients who may be requiring a higher level of care. This system enables both nurses and physicians to notify the RRT and have a critical care team evaluate the patients. During the period of 03/01/2018 to 09/17/2018, Mount Sinai Hospital floor units on 10W and 10E units made 357 rapid response team (RRT) calls with only 58 leading to an actual increase in the level of care (true positive rate ~ 16%). Similarly, the Electronic Health Record (EHR) generated 839 sepsis Best Practice Alerts (BPAs) yet only five led to escalations in care (true positive rate ~ 0.5%). The results above would imply that over 168 evaluations need to be made to identify a single case where the patient required an escalation in care. The goal of ReSCUE-ME is to evaluate prospective model performance and identify the best spot which the study team can incorporate MEWS++ into RRT and Primary providers workflow. The primary endpoint is rate of escalation of care on 10W and 10E during the study period.

Background:

In a prior study, the group has demonstrated that a machine learning model (MEWS++) significantly outperformed a standard, manually calculated MEWS score on a large retrospective cohort of hospitalized patients. To develop this model, the study team used a data set (Approved by the Program for Protection of Human Subjects Institutional Review Board (IRB) IRB-18-00581) of 96,645 patients with 157,984 hospital encounters and 244,343 bed movements. The study team found that MEWS++ was superior to the standard MEWS model with a sensitivity of 81.6% vs. 44.6%, specificity of 75.5% vs. 64.5%, and area under the receiver operating curve of 0.85 vs. 0.71.

Encouraged by this prior result, the study team is seeking to evaluate the model in a prospective study.

A silent pilot of the ReSCUE-ME alerts has been running on 10E and 10W since Feb 2019. The study team has continuously monitoring the alert performance via a real-time web-based dashboard. The results are summarized below:

* Median # of alerts to primary team, per floor, per day: 8
* Median # of alerts to RRT, per floor, per day: 4
* Sensitivity 0.76, Specificity 0.68, AUC 0.77
* Accuracy 0.69, Precision 0.3, F1 Score 0.43 This performance compares very favorably to the performance seen in the retrospective historical cohort used to develop the MEWS++ model:
* Sensitivity 0.82, Specificity 0.76, AUC 0.85
* Accuracy 0.76, Precision 0.12, F1 Score 0.19"

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18 or greater who were admitted to a general care unit selected for each arm.

Exclusion Criteria:

* Any admitted patient who has a "Do Not Resuscitate (DNR)" and/or a "Do Not Intubate (DNI)" order in the EHR,
* any patient made "level of care" by RRT as documented in REDCap.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2780 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Levin, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified raw data may be shared with other researchers upon submission of a written request along with a plan for how the data are intended to be used.

REFERENCES:
- [Derived] Levin MA, Kia A, Timsina P, Cheng FY, Nguyen KA, Kohli-Seth R, Lin HM, Ouyang Y, Freeman R, Reich DL. Real-Time Machine Learning Alerts to Prevent Escalation of Care: A Nonrandomized Clustered Pragmatic Clinical Trial. Crit Care Med. 2024 Jul 1;52(7):1007-1020. doi: 10.1097/CCM.0000000000006243. Epub 2024 Feb 21. PMID 38380992

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients admitted to the study units were enrolled. There were no opt-outs.
Period: Overall Study
Arm/Group | MEWS++ Monitoring | Standard of Care Monitoring
Started | 1506 | 1274
Completed | 1506 | 1274
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MEWS++ Monitoring | Standard of Care Monitoring | Total
Number analyzed (Participants) | 1488 | 1252 | 2740
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (17) | 65.1 (17.8) | 66.2 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 762 | 666 | 1428
  Male | 726 | 586 | 1312
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 472 | 433 | 905
  Not Hispanic or Latino | 1016 | 819 | 1835
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 541 | 401 | 942
  Black | 367 | 287 | 654
  Asian | 83 | 94 | 177
  Other | 480 | 448 | 928
  Missing | 17 | 22 | 39
BMI [Mean (Standard Deviation); unit: kg per meters squared] | 27.1 (7.68) | 26.5 (9.1) | 26.9 (8.34)
Elixhauser Score [Mean (Standard Deviation); unit: units on a scale] — A measure of the overall severity of comorbidities, based on ICD diagnosis codes. Range is -19 to +89, with a score of > +15 indicating severe comorbid illness.
  units on a scale | 2.2 (1.4) | 2.2 (1.4) | 2.2 (1.4)
First Deterioration Score on Admission [Mean (Standard Deviation); unit: proportion probability] — Predicted likelihood of escalation to intensive care or death in hospital. This score is the output of the MEWS++ random forest model. Data from the EHR, laboratory information system and ECG system were used. Features included laboratory test results, vital signs, automated ECG interpretations, and structured clinical nursing documentation (e.g., level of consciousness). Full model description published in PMID 32012659. Range 0-1. Cutoff for a positive prediction 0.59. At this threshold the sensitivity was 0.4, specificity 0.78, PPV 0.13, and NPV 0.94 for ICU escalation or death.
  proportion probability | 0.56 (0.1) | 0.57 (0.096) | 0.57 (0.098)

OUTCOME MEASURES:

1. Primary Outcome: Overall Rate of Escalation
Description: Rate of escalation of care from floor to Stepdown, Telemetry, ICU, per 1,000 patient bed days.
Time Frame: 10 months
Measure: Number; unit: escalations per 1,000 patient bed days
Groups:
- Intervention - Alert Sent: A score predicting the likelihood that the patient will experience a deterioration in their clinical condition within six hours will be generated. If the prediction score exceeds a predetermined threshold, an alert will be sent to the provider. The alerting protocol is tiered, with both a low and high threshold. If the score is above the low threshold, nursing will be notified. If the score is above the high threshold, RRT will be notified.
- Control - Standard of Care Monitoring: A score predicting the likelihood that the patient will experience a deterioration in their clinical condition within six hours will be generated.Patients in the control arm will have a score calculated but no alert will be sent.
Arm/Group | Intervention - Alert Sent | Control - Standard of Care Monitoring
Number analyzed (Participants) | 1488 | 1252
escalations per 1,000 patient bed days | 12.3 | 11.3
Statistical Analysis 1: Comparison: Intervention - Alert Sent vs Control - Standard of Care Monitoring; IPTW Poisson regression was used to model the number of escalations per visit with an offset of the log transformed length of stay normalized per 1000 bed days. Treatment effect is expressed in terms of adjusted incidence rate ratio (IRR) per 1000 patient bed days; Test type: Superiority; p < 0.001, Regression, Poisson; Risk Ratio (RR) = 1.43, 95% CI 2-sided [1.16 to 1.78]

2. Secondary Outcome: Number of Participants Requiring Blood Pressure Support
Description: Number of participants requiring blood pressure support agents such as initiation of vasopressor medication or administration of fluid bolus.
Time Frame: 10 months
Measure: Count of Participants; unit: Participants
Groups:
- Control - No Alert Sent: A score predicting the likelihood that the patient will experience a deterioration in their clinical condition within six hours will be generated. Patients in the control arm will have a score calculated but no alert will be sent.
Arm/Group | Intervention - Alert Sent | Control - No Alert Sent
Number analyzed (Participants) | 1488 | 1252
Participants | 239 | 142
Statistical Analysis 1: Comparison: Intervention - Alert Sent vs Control - No Alert Sent; IPTW log-binomial regres- sion models were used to model the secondary and ad hoc outcomes. Treatment effect is expressed as adjusted relative risk (RR); Test type: Superiority; p < 0.001, Regression, Logistic — Correction for multiple comparisons was performed on all key outcomes within the primary and secondary hypotheses, respectively, using the false discovery rate method (FDR); Risk Ratio (RR) = 1.74, 95% CI 2-sided [1.39 to 2.18]

3. Secondary Outcome: Number of Participants Requiring Respiratory Support
Description: Number of participants requiring respiratory support intervention such as initiation of nasal cannula to high flow or frequency of intubation.
Time Frame: 10 months
Population: No statistical comparison performed due to low rate of events.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention - Alert Sent | Control - No Alert Sent
Number analyzed (Participants) | 1488 | 1252
Participants | 15 | 5

4. Secondary Outcome: Number of Participants Who Experienced a Cardiac Arrest Episode
Description: The number of patients who had a cardiac arrest.
Time Frame: 10 months
Population: No statistical comparison performed due to no events.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention - Alert Sent: A score predicting the likelihood that the patient will experience a deterioration in their clinical condition within six hours will be generated. If the prediction score exceeds a predetermined threshold, an alert will be sent to the provider.
Arm/Group | Intervention - Alert Sent | Control - No Alert Sent
Number analyzed (Participants) | 1488 | 1252
Participants | 0 | 0

5. Secondary Outcome: Mortality Rate
Description: Number of Mortalities - Combined In-hospital and 30-day mortality. Mortalities only counted once. 30-day mortality includes those patients who died in-hospital within 30 days.
Time Frame: Duration of hospital stay, until discharge, regardless of stay length for patients who died in hospital, or 30 days after admission, starting from date of admission, up to 6 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention - Alert Sent | Control - No Alert Sent
Number analyzed (Participants) | 1488 | 1252
Participants
  Combined in-hospital and 30-day | 104 | 117
  In-hospital mortality | 81 | 83
  30-d mortality | 87 | 98
Statistical Analysis 1: Comparison: Intervention - Alert Sent vs Control - No Alert Sent; IPTW log-binomial regression models were used to model the secondary and ad hoc outcomes. Treatment effect is expressed as adjusted relative risk (RR); Test type: Superiority; p = 0.045, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 0.76, 95% CI 2-sided [0.58 to 0.99]

6. Secondary Outcome: Notification Frequency - Number of Alerts Sent Per Day to Providers
Description: The number is calculated as average number of alerts sent per day over all the days in the study period.
Time Frame: 10 months
Population: No statistical analysis performed
Measure: Mean (Standard Deviation); unit: alerts per day
Arm/Group | Intervention - Alert Sent | Control - No Alert Sent
Number analyzed (Participants) | 1488 | 1252
alerts per day
  Total Alerts | 6.7 (3.0) | 5.4 (2.5)
  Primary Alerts | 4.5 (2.3) | 3.5 (1.9)
  RRT Alerts | 2.2 (1.7) | 1.9 (1.5)

7. Secondary Outcome: Number of Calls
Description: The average number of calls to RRT made per patient, regardless of alert. Not evaluated.
Time Frame: 10 months
Population: Data were not collected for this outcome measure.
Arm/Group | Intervention - Alert Sent | Control - Standard of Care Monitoring
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Sensitivity and Specificity of the RRT Alert
Description: The performance of the alert will be evaluated by calculating the sensitivity, specificity, positive predictive value, negative predictive value, precision, recall, and F1-score. This will be done both for the overall escalation rate and if possible for individual escalations (ICU, step-down, telemetry) and death.
Time Frame: 10 months
Population: Patients in the intervention arm.
Measure: Number; unit: proportion
Arm/Group | Intervention - Alert Sent
Number analyzed (Participants) | 1506
proportion
  Sensitivity | 0.88
  Specificity | 0.33
  Positive Predictive Value | 0.15
  Negative Predictive Value | 0.95

9. Post Hoc Outcome: Time to ICU Escalation
Description: Time in hours between alert and transfer to an ICU
Time Frame: From time of alert until transfer to an ICU, assessed up to discharge from the hospital or death
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Intervention - Alert Sent | Control - No Alert Sent
Number analyzed (Participants) | 1488 | 1252
hours | 49.7 [21.6 to 101] | 57.8 [25.2 to 113]

10. Post Hoc Outcome: Likelihood of Earlier Hospital Discharge
Description: Hazard ratio for faster earlier discharge for patients who got an alert
Time Frame: Duration of hospital stay, starting from admission, up to the day of discharge, regardless of the length of hospital stay, up to 1 year.
Population: Patients who survived to hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention - Alert Sent | Control - Standard of Care Monitoring
Number analyzed (Participants) | 1488 | 1252
Participants | 1407 | 1,169
Statistical Analysis 1: Comparison: Control - Standard of Care Monitoring; Test type: Superiority; p = 0.14, Regression, Cox; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.98 to 1.18]

ADVERSE EVENTS:
Time Frame: All-cause mortality data were collected up to 30 days post-admission from hospital, up to 6 weeks post-admission.
Description: No adverse event data were collected other than all cause mortality.
Arm/Group | MEWS++ Monitoring | Standard of Care Monitoring
All-Cause Mortality (participants affected / at risk) | 104/1488 | 117/1252
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT04026555/Prot_SAP_000.pdf